CLINICAL TRIAL: NCT06645028
Title: Evaluation of an 8-day Intensive Treatment Programme for PTSD and CPTSD in the Swedish Mental Health Care
Brief Title: 8-day Intensive Treatment Programme for PTSD and CPTSD in Sweden
Acronym: 8-day ITP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Blomdahl (Other Government)
Collaborators: Vastra Gotaland Region (Other Government); Sodra Alvsborgs Hospital (Other)
Responsible Party: Sponsor-Investigator, Christina Blomdahl, R & D Strategic, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 280348
Record Dates: First submitted 2024-09-20; First posted 2024-10-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-10

CONDITIONS: PTSD; Complex Post-Traumatic Stress Disorder
Keywords: Intensive treatment programme; EMDR; Prolonged exposure; Physical activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Intervention Model Description: Open clinical trail where participants are allocated via shared desicion making
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive treatment programme (Experimental): Intervention Group: 8-day intensive treatment where each treatment day consists of the following schedule: Physical activity: 30 minutes Prolonged Exposure (PE): 90 minutes Physical activity: 30 minutes Lunch Physical activity: 60 minutes Eye Movement Desensitization and Reprocessing (EMDR): 90 minutes Physical activity: 30 minutes (omitted on days 4 and 8) Dinner Psychoeducation (omitted on days 4 and 8) Participants stay at the SÄS patient hotel during the treatment (with a three-day weekend break between treatment days 1-4 and 5-8). The treatment concept includes therapist rotation, meaning that participants switch therapists between PE and EMDR sessions. The purpose of this is to increase focus on the processing process rather than the relationship between the therapist and the client.
  Interventions: Behavioral: Intensive treatment programme
- Treatment as usual (Active Comparator): Control group: 16 treatment sessions (90 minutes in duration) either Eye movement desensitisation and reprocessing (EMDR) or Prolonged Exposure (PE) in a standard outpatient format-weekly sessions. Participants can choose to attend 6 sessions of Psychoeducation for PTSD in a group format before starting EMDR or PE.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Intensive treatment programme — Intervention Group: 8-day intensive treatment where each treatment day consists of the following schedule:
  Physical activity: 30 minutes Prolonged Exposure (PE): 90 minutes Physical activity: 30 minutes Lunch Physical activity: 60 minutes Eye Movement Desensitization and Reprocessing (EMDR): 90 minutes Physical activity: 30 minutes (omitted on days 4 and 8) Dinner Psychoeducation (omitted on days 4 and 8) Participants stay at the SÄS patient hotel during the treatment (with a three-day weekend break between treatment days 1-4 and 5-8). The treatment concept includes therapist rotation, meaning that participants switch therapists between PE and EMDR sessions. The purpose of this is to increase focus on the processing process rather than the relationship between the therapist and the client.
  Other Names: EMDR; Prolonged Exposure
  Arms: Intensive treatment programme
Behavioral: Treatment as Usual (TAU) — Control group: 16 treatment sessions (90 minutes in duration) either Eye movement desensitisation and reprocessing (EMDR) or Prolonged Exposure (PE) in a standard outpatient format-weekly sessions. Participants can choose to attend 6 sessions of Psychoeducation for PTSD in a group format before starting EMDR or PE.
  Other Names: Prolonged Exposure; EMDR
  Arms: Treatment as usual

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) and Complex PTSD (C-PTSD) are conditions that may develop after a person has been exposed to extremely stressful experiences. The affected individual re-experiences the event despite attempts to avoid reminders of the experience and also experiences heightened tension. In C-PTSD, the individual also experiences significantly impaired ability to regulate emotions, severe negative change in self-image, and difficulty maintaining close relationships.

Traditional trauma-focused psychotherapy for PTSD typically involves one session per week over approximately 6-12 months. Intensive treatment models for both PTSD and C-PTSD have been developed and have shown promising results, with lower dropout rate from treatment compared to traditional treatments. The current project aims to compare the outcomes of an 8-day intensive treatment programme with treatment in a traditional format. Individuals with C-PTSD or PTSD who have not benefited from previous treatment attempts are included in the study. Participants are allocated to the respective treatment group according to principles of person-centered care, where participants are considered competent to make an informed choice of treatment method.

Diagnostic assessment and self-rating of symptoms of PTSD and C-PTSD are conducted before and after treatment, as well as at 3-month follow-up. The study is expected to provide increased knowledge on whether 8-day intensive treatment is a suitable alternative to treatment in a traditional format for PTSD and C-PTSD. The study is also expected to provide important data for considering whether 8-day intensive treatment should be widely implemented in Swedish psychiatry.

DETAILED DESCRIPTION:
1. Study aims and research questions

   The purpose of the study is to compare the outcomes and potential risks between two treatment methods for treatment-resistant PTSD and C-PTSD: 8-day intensive treatment and conventional treatment. Additionally, the study aims to investigate whether there are individual factors that influence the outcomes of each treatment format.

   Specific research questions:

   • Can a difference in the severity of PTSD and C-PTSD be observed after 8-day intensive treatment? Does the outcome differ compared to conventional treatment for PTSD and C-PTSD?

   • Are there individual factors that influence the treatment outcome? Does the impact of these factors differ between the study groups?

   • Does participation in 8-day intensive treatment pose an increased risk of adverse, harmful effects or an increase in suicidal intentions during and after the treatment?
2. Method

2.1 Participants

Participants consist of individuals referred to the Adult Psychiatric Outpatient Clinic for Psychosis and PTSD at Södra Älvsborgs Hospital between August 2021 and December 2023. Inclusion criteria for participation: diagnosis of C-PTSD or PTSD with previous treatment attempts that have not been effective. Exclusion criteria: insufficient knowledge of the Swedish language to respond to questionnaires, need for an interpreter during treatment, use of benzodiazepines, acute suicidality, or dissociative identity disorder. All individuals who meet the inclusion criteria during the recruitment period are asked about their willingness to participate.

We calculated differences between two independent groups with means. The calculation was based on the PCL-5 and the results from the study by Wortmann et al. (2016). The power calculation was performed using G*Power 3.1.9.4 (Faul et al., 2007) With a power of 0.80, a significance level of 0.05, a two-sided test, Group 1 had a difference of 10 (SD 15), and Group 2 had a difference of 2 (SD 13). The effect size was 0.56, which corresponds to a moderate effect. This results in a total sample of 100, i.e., 50 participants in each group.

2.2 Procedure

Allocation to each intervention group follows the principles of person-centered care, where participants are considered competent to be involved in their treatment choice. Participants are provided with written and verbal information about the treatment options and given the opportunity to ask questions in order to make an informed decision.

2.3 Data collection

Data is collected in the two following ways:

1. Through questionnaires and clinician ratings conducted during the inclusion assessment and follow-up after treatment, the following data is collected:

   • Trauma history (LEC-5),

   • Diagnosis of PTSD or C-PTSD (ITI 3.2),
   * Self-assessment of dissociative symptoms (DES II),
   * Clinician rating of suicidal intentions (SSI).
2. Data is collected via the REDcap database before, during, and after treatment completion. Participants receive a printed QR code for each assessment point and complete the assessments via mobile phone or computer. If needed, assessments can be done manually. The digital assessments include:

   * Background information such as demographic data, sick leave status, employment, psychiatric treatment history, and ongoing treatment.
   * Self-report questionnaires measuring PTSD symptoms (PCL-5), C-PTSD symptoms (ITQ), and transdiagnostic screening of psychiatric symptoms (DSM-5 CCM Level 1).

2.4. Data analysis

Analysis of group differences and exploratory analyses will be conducted using statistical software (SPSS for Windows). Differences in background data and baseline data between groups will be tested using the Chi-square (X²) test for categorical data and independent t-tests for numerical data, or alternatively, the Mann-Whitney U test if the criteria for parametric statistics are not met for numerical data.

* Data from all included participants completing basline assessment will be used, regardless of the number of completed assessments. Data that are possible statistical outliers will be included in the analysis if they are not outside the expected clinical range for the specific measure. Intent-to-treat (ITT) analysis will be applied to analyze outcomes related to repeated measurements (PCL-5 and ITQ). For this purpose, Linear Mixed Model (LMM) will be used, allowing for the inclusion of all available data from participants across all time points.

  - Difference between groups will be analyzed for means and standard deviations. Results will be presented with levels of signifiance (p.05) and effectsize, including confidence intervals.
* Exploratory analysis of moderating individual factors (baseline symptom measurement, demographics, comorbidity, trauma history) that may influence treatment outcomes will be conducted using multiple regression analysis.

  3. Expected outcomes and contributions fot the field of knowledge

The study is expected to provide increased knowledge on whether 8-day intensive treatment has an impact on symptoms in treatment-resistant forms of PTSD and C-PTSD, and whether its effectiveness differs from traditional treatment. The study is also anticipated to enhance understanding of whether individual factors play a role in the choice of treatment.

Overall, the study aims to provide important insights into intensive treatment for C-PTSD and treatment-resistant PTSD in a Swedish context. This knowledge is expected to contribute to decisions on whether intensive treatment should be implemented in Swedish psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* CPTSD according to ICD-11
* PTSD with at least one comorbid disorder requiring psychiatric outpatient treatment
* PTSD with previous unsuccessful trauma-focused treatment

Exclusion Criteria:

* ongoing substance or alcohol abuse
* use of benzodiazepines
* acute suicidality
* dissociative identity disorder (DID)
* insufficient knowledge of the Swedish language to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Checklist for DSM-5 (PCL-5) | Pre-treatment: 2 weeks before start. Posttreatment: 1 week after treatment. Follow-up: 3 months after treatment. Repeated measure at session 2,4,6,8,10,12,14. In ITP this corresponds to day 1-7 of treatment. TAU this corresponds to week 2-14 of treatm.
  Self-report measure of PTSD symptoms according to DSM-5 criteria. PCL-5 contains 20 items, rated on a 5-point scale (0 = "not at all" to 4 ("extremely"). It has shown good internal reliability (.96) and test-retest reliability (.84) (Bovin et al., 2016). PCL-5 has also demonstrated sensitivity to clinical change during treatment (Marx et al., 2022)

SECONDARY OUTCOMES:
International Trauma Questionnaire (ITQ) | Pre-treatment: 2 weeks before start. Posttreatment: 1 week after treatment. Follow-up: 3 months after treatment.
  A self-report measure developed to measure PTSD symptoms and C-PTSD symptoms according to ICD-11. ITQ contains 18 items in total, 12 items to asses symptoms (6 for PTSD and 6 for PTSD) and six items to assess functional disability associated with PTSD and C-PTSD. In this study, only items measuring symptoms were included. Items are rated on a 5-point Likert scale (0 = "not at all" to 4 ("extremely"). ITQ has shown good internal reliability (.89 to .94) (Cloitre et al., 2021).

OTHER OUTCOMES:
International Trauma Interview (ITI) 3.2 (test version) | Pre-treatment: 2 weeks before start. Posttreatment: 1 week after treatment. Follow-up: 3 months after treatment.
  For diagnostic assessment of PTSD and CPTSD, the International Trauma Interview (ITI) 3.2 (test version) (Roberts, 2019) was used. ITI 3.2 is an interview divided into two parts. Part one has 7 items to help the interviewer assess the three symptom domains of PTSD (re-experiencing, avoidance, hyperarousal) and 2 items to assess functional disability. Part 2 has 6 items to assess the three DSO domains (affect regulation, self-image, relationship difficulties), and 2 items to assess functional disability. All items are evaluated on a 5-point scale, based on symptom intensity and frequency during the last month (0 = "absent" to 4 = "extremely). Ratings are summoned in a matrix where at least one item per symptom domain must be rated ≥2, and at least one item for functional disability must be rated ≥ 2 to make up a diagnosis of PTSD and C-PTSD (PTSD + DSO), respectively. In the study ITI was used to assess PTSD and C-PTSD on a categorical level (diagnosis or no diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Blomdahl, PhD, Principal Investigator — REDI, Primary Health Care, Västra Götalands Region (VGR); Sandra Weineland, Associate Professor, Study Director — Dpt of Psychology, Gothenburg University; REDI, Primary Health Care, VGR
Locations (1):
- Södra Älvsborgs Sjukhus, Västra Götalandsregion, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No
Under the rules of General Data Protection Regulation, GDPR, sharing of sensitive data regarding individuals is regulated. Careful assessment of whether individuals can be identified via IPD before decision on sharing of data can be made.

REFERENCES:
- [Background] Van Woudenberg C, Voorendonk EM, Bongaerts H, Zoet HA, Verhagen M, Lee CW, van Minnen A, De Jongh A. Effectiveness of an intensive treatment programme combining prolonged exposure and eye movement desensitization and reprocessing for severe post-traumatic stress disorder. Eur J Psychotraumatol. 2018 Jul 10;9(1):1487225. doi: 10.1080/20008198.2018.1487225. eCollection 2018. PMID 30013726
- [Background] Sciarrino NA, Warnecke AJ, Teng EJ. A Systematic Review of Intensive Empirically Supported Treatments for Posttraumatic Stress Disorder. J Trauma Stress. 2020 Aug;33(4):443-454. doi: 10.1002/jts.22556. Epub 2020 Jun 29. PMID 32598561
- [Background] Voorendonk EM, De Jongh A, Rozendaal L, Van Minnen A. Trauma-focused treatment outcome for complex PTSD patients: results of an intensive treatment programme. Eur J Psychotraumatol. 2020 Jul 23;11(1):1783955. doi: 10.1080/20008198.2020.1783955. PMID 33029323
- See also: Description of the project in Swedish — https://www.researchweb.org/is/se/vgr/project/280348